CLINICAL TRIAL: NCT02876107
Title: A Randomized Phase II Study of Neoadjuvant Carboplatin/Paclitaxel (CT) Versus Panitumumab/Carboplatin/Paclitaxel (PaCT) Followed by Anthracycline-Containing Regimen for Newly Diagnosed Primary Triple-Negative Inflammatory Breast Cancer
Brief Title: Carboplatin and Paclitaxel With or Without Panitumumab in Treating Patients With Invasive Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0177; NCI-2017-00619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0177 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma; Breast Lump; Edema; Erythema; Estrogen Receptor Negative; HER2/Neu Negative; Inflammatory Breast Carcinoma; Invasive Breast Carcinoma; Peau d'Orange; Progesterone Receptor Negative; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Edema; Erythema; Inflammatory Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (panitumumab, paclitaxel, carboplatin) (Experimental): Patients receive panitumumab IV over 1 hour on day 1 of cycle 0 and over 30 minutes on days 1, 8, and 15 of cycles 1-4. Patients also receive paclitaxel IV over 1-3 hours on days 1, 8, and 15 of cycles 1-4, and carboplatin IV over 30 minutes on day 1 of cycles 1-4. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Panitumumab
- Group B (paclitaxel, carboplatin) (Experimental): Patients receive paclitaxel, carboplatin, doxorubicin, and cyclophosphamide as in Group A. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix
  Arms: Group A (panitumumab, paclitaxel, carboplatin)

SUMMARY:
This randomized phase II trial studies how well carboplatin and paclitaxel with or without panitumumab work in treating patients with invasive triple negative breast cancer. Drugs used in the chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping the them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as panitumumab, may interfere with the ability of tumor cells to grow and spread. Giving carboplatin and paclitaxel with or without panitumumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pathologic complete response (pCR) rate in patients with primary triple-receptor negative (estrogen receptor [ER]-negative, progesterone receptor [PgR]-negative, and human epidermal growth factor receptor 2 [HER2]-negative) inflammatory breast cancer (TN-IBC) by using a combination of panitumumab, carboplatin, and paclitaxel (PaCT) in comparison with carboplatin and paclitaxel (CT) followed by adriamycin and cyclophosphamide (AC) in a neoadjuvant setting.

SECONDARY OBJECTIVES:

I. To determine the disease-free survival (DFS) rates produced by either arm of trial combination treatment.

II. To determine the overall survival (OS) rates produced by either arm of trial combination treatment.

III. To determine the safety and tolerability of both arms of trial combination treatment.

EXPLORATORY OBJECTIVES:

I. To determine whether the pCR rate positively correlates with reduced nodal expression status.

II. To determine whether the pCR rate inversely correlates with arginine methylation status of epidermal growth factor receptor (EGFR).

III. To identify molecular biomarkers predictive of the pCR rate by analysis of multiplexed immunohistochemical (IHC) staining.

IV. To identify molecular biomarkers predictive of the pCR rate by genomic and proteomic analysis.

V. To determine whether the inhibition of the EGFR pathway downregulates the COX-2 pathway and mesenchymal marker.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP A: Patients receive panitumumab intravenously (IV) over 1 hour on day 1 of cycle 0 and over 30 minutes on days 1, 8, and 15 of cycles 1-4. Patients also receive paclitaxel IV over 1-3 hours on days 1, 8, and 15 of cycles 1-4, and carboplatin IV over 30 minutes on day 1 of cycles 1-4. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unexpected toxicity.

GROUP B: Patients receive paclitaxel, carboplatin, doxorubicin, and cyclophosphamide as in Group A. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up at 1 month and then annually for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological confirmation of breast carcinoma
* Patients must have invasive breast cancer (IBC), confirmed according to international consensus criteria:

  * Onset: Rapid onset of breast erythema, edema, and/or peau d'orange, and/or warm breast, with or without an underlying breast mass
  * Duration: History of such findings no more than 6 months
  * Extent: Erythema occupying at least 1/3 of whole breast
  * Pathology: Pathologic confirmation of invasive carcinoma
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must have negative HER2 expression on immunohistochemistry (IHC) (defined as 0 or 1+) or fluorescence in situ hybridization (FISH) analysis; if HER2 is 2+, negative HER2 expression must be confirmed by FISH (HER2/cep17 ration < 2, and/or copy number less than 6); ER and PgR expression should be less than 10%
* Patients have left ventricular ejection fraction (LVEF) >= 50% by multigated acquisition scan (MUGA) or echocardiogram before study randomization
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Hemoglobin >= 9.0 g/dL
* Aspartate aminotransferase (AST) =< 3.0 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) =< 3.0 x ULN
* Alkaline phosphatase (ALP) =< 2.5 x ULN
* Total bilirubin =< 1.5 x ULN
* Creatinine (Cr) =< 1.5 mg/dL x ULN
* Creatinine clearance (CrCl) >= 50 mL/min calculated by the Cockroft-Gault
* Patients have the ability and willingness to sign written informed consent
* Patients of childbearing potential (women who are postmenopausal for < 1 year, not surgically sterilized, or not abstinent), have a negative urine pregnancy test, and agree to the consistent and correct use of one of the following acceptable methods of birth control: male partner who is sterile before the female subject's entry into the study and is the sole sexual partner for that female subject; intrauterine device, oral contraception, or barrier methods, including diaphragm or condom with a spermicide

Exclusion Criteria:

* Stage IV disease, if the metastatic sites are not amendable for local therapy (i.e. radiation and/or surgery), and are not candidates for breast surgery will not be eligible
* History of radiotherapy for current breast cancer diagnosis
* History of recent malignancies < 5 years (except for cured non-melanomatous skin cancer or cured cervical carcinoma in situ)
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, acute or chronic active hepatitis B infection
* History of extensive interstitial lung disease, e.g., pneumonitis or pulmonary fibrosis or any evidence of extensive interstitial lung disease on baseline chest computed tomography (CT) scan
* Other known other significant medical or psychiatric condition that would make assessment of toxicity or efficacy difficult
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a peripheral neuropathy > grade 1
* Patients with a history of New York Heart Association class 3 or 4 heart failure, or history of myocardial infarction, unstable angina, or cerebrovascular accident (CVA) within 6 months of protocol registration
* Patients have a history of prior therapy with carboplatin
* Patients have received a cumulative dose of doxorubicin of greater than 360 mg/m^2 or epirubicin of greater than 640 mg/m^2
* Patients have had prior radiotherapy for primary breast carcinoma or axillary lymph nodes
* Patients have history of diagnosed interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Complete pathologic response | At the time of surgery, assessed up to 5 years
  Will be estimated for each treatment arm with exact 95% confidence intervals. A Chi-square test or Fisher's exact test will be used to compare the differences in complete pathologic response rate between the two treatment arms. A logistic regression model will be used to assess the differences in complete pathologic response between the two treatment arms, adjusting for other covariates as appropriate. The analysis will be based on the modified intent-to-treat population.

SECONDARY OUTCOMES:
Disease free survival | Up to 5 years
  The method of Kaplan-Meier method will be used to estimate the time-to-event outcomes.
Overall survival | Up to 5 years
  The method of Kaplan-Meier method will be used to estimate the time-to-event outcomes.
Incidence of adverse events | Up to 5 years
  Descriptive statistics will be used.

OTHER OUTCOMES:
Reduced nodal expression status | Up to 5 years
  Descriptive statistics will be summarized for all the variables collected in this study. For continuous variables, mean, standard deviation, median, and range will be presented. For categorical variables, frequency tables will be provided. To compare the continuous variables between/among groups, either the parametric method (two-sample t-test or analysis of variance method) or nonparametric method (Wilcoxon or Kruskal-Wallis test) will be used, depending on the distribution of the data. For testing correlation between two categorical variables, either the Chi-square test or Fisher's exact test will be used.
Arginine methylation status of EGFR | Up to 5 years
  Descriptive statistics will be summarized for all the variables collected in this study. For continuous variables, mean, standard deviation, median, and range will be presented. For categorical variables, frequency tables will be provided. To compare the continuous variables between/among groups, either the parametric method (two-sample t-test or analysis of variance method) or nonparametric method (Wilcoxon or Kruskal-Wallis test) will be used, depending on the distribution of the data. For testing correlation between two categorical variables, either the Chi-square test or Fisher's exact test will be used.
Molecular biomarkers assessed by genomic and proteomic analysis | Up to 5 years
  Descriptive statistics will be summarized for all the variables collected in this study. For continuous variables, mean, standard deviation, median, and range will be presented. For categorical variables, frequency tables will be provided. To compare the continuous variables between/among groups, either the parametric method (two-sample t-test or analysis of variance method) or nonparametric method (Wilcoxon or Kruskal-Wallis test) will be used, depending on the distribution of the data. For testing correlation between two categorical variables, either the Chi-square test or Fisher's exact test will be used.
Downregulation of COX-2 pathway and mesenchymal marker by EGFR pathway | Up to 5 years
  Descriptive statistics will be summarized for all the variables collected in this study. For continuous variables, mean, standard deviation, median, and range will be presented. For categorical variables, frequency tables will be provided. To compare the continuous variables between/among groups, either the parametric method (two-sample t-test or analysis of variance method) or nonparametric method (Wilcoxon or Kruskal-Wallis test) will be used, depending on the distribution of the data. For testing correlation between two categorical variables, either the Chi-square test or Fisher's exact test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Nasrazadani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wang X, Zhao L, Song X, Wu X, Krishnamurthy S, Semba T, Shao S, Knafl M, Coffer LW 2nd, Alexander A, Vines A, Bopparaju S, Woodward WA, Chu R, Zhang J, Yam C, Loo LWM, Nasrazadani A, Huong LP, Woodman SE, Futreal A; Rare Tumor Initiative Team; Tripathy D, Ueno NT. Genomic and transcriptomic analyses identify distinctive features of triple-negative inflammatory breast cancer. NPJ Precis Oncol. 2024 Nov 18;8(1):265. doi: 10.1038/s41698-024-00729-0. PMID 39558017
- See also: MD Anderson Cancer Center — http://www.mdanderson.org